CLINICAL TRIAL: NCT05381012
Title: The Effect of Fibromyalgia Syndrome on Female Patients With Chronic Migraine
Brief Title: Fibromyalgia Syndrome on Patients With Chronic Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Alper mengi, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 26.04.2022/372690
Record Dates: First submitted 2022-05-14; First posted 2022-05-19 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Chronic Migraine, Headache; Fibromyalgia Syndrome; Chronic Pain Syndrome; Central Sensitisation; Headache Disorders
MeSH Terms: conditions — Headache; Fibromyalgia; Headache Disorders | interventions — Quality of Life; Sleep; Central Nervous System Sensitization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronic migraine (Other): Patients diagnosed with chronic migraine according to the International Headache Society Classification (ICHD-3).
  Interventions: Other: Allodynia, quality of life, sleep, anxiety and depression, disability, and central sensitization
- Fibromyalgia syndrome (Other): Patients diagnosed with chronic migraine according to the International Headache Society Classification (ICHD-3), and patients with fibromyalgia syndrome .
  Interventions: Other: Allodynia, quality of life, sleep, anxiety and depression, disability, and central sensitization; Other: Fibromyalgia syndrome

INTERVENTIONS:
Other: Allodynia, quality of life, sleep, anxiety and depression, disability, and central sensitization — All patients will be evaluated for allodynia, quality of life, sleep, anxiety and depression, disability related to headache, and central sensitization.
Other: Fibromyalgia syndrome — Patients who meet the diagnostic criteria for fibromyalgia syndrome will be evaluated with the Fibromyalgia Impact Questionnaire.
  Arms: Fibromyalgia syndrome

SUMMARY:
The aim of this study to evaluate the effects of fibromyalgia syndrome accompanying women with chronic migraine on pain, quality of life, sleep, anxiety and depression, central sensitization and functionality.

DETAILED DESCRIPTION:
Patients who applied to Istanbul University-Cerrahpaşa, Cerrahpaşa Faculty of Medicine, Department of Neurology, headache outpatient clinic and were diagnosed with chronic migraine according to the International Headache Society Classification (ICHD-3), after the patient's history and physical examination, will be included in the study.

Date of birth, education level, body mass index, occupation, marital status, socioeconomic status, age of onset of migraine complaints, descriptive information about migraine attacks (type (with or without aura), duration of attacks, average number of days with pain, pain severity, accompaniments) will be questioned.

In addition, if the fibromyalgia syndrome meets the diagnostic criteria, symptom duration and average body pain severity in the last 3 months will be questioned.

A total of 66 patients are planned to be included in the study. In the study, 2 groups will be formed, the first group will consist of chronic migraine patients, the second group will consist of patients with chronic migraine as well as fibromyalgia syndrome.

All patients will be evaluated for allodynia, quality of life, sleep, anxiety and depression, disability related to headache, and central sensitization. Relevant forms will be filled by patients.

Patients will be evaluated with the diagnostic criteria for fibromyalgia syndrome and if the patients meet the diagnostic criteria for fibromyalgia syndrome, the Fibromyalgia Impact Questionnaire will be applied. The patient will be evaluated by Alper Mengi in terms of fibromyalgia syndrome diagnostic criteria.

ELIGIBILITY:
Inclusion Criteria:

For patients with chronic migraine:

* Being diagnosed with chronic migraine according to the International Headache Society Classification (ICHD-3)
* Being literate

For patients with fibromyalgia syndrome:

* Diagnosed with chronic migraine according to the International Headache Society Classification (ICHD-3)
* Being literate
* Diagnosed with fibromyalgia syndrome according to the 2016 American College of Rheumatology criteria

Exclusion Criteria:

* Having another pathology that can explain their pain in the head and face region other than chronic migraine (such as sinusitis, tension-type headache, trigeminal neuralgia, drug overuse headache)
* Psychiatric disease or using psychiatric drugs
* History of serious head trauma or neurosurgical intervention
* History of infectious, chronic inflammatory disease, malignancy
* Pregnant and breastfeeding women
* History of additional neurological disease other than migraine
* Uncooperative
* Having congestive heart failure, chronic kidney failure, chronic liver disease, lung disease, uncontrolled diabetes, peripheral vascular disease
* Diagnosed with hypothyroidism or hyperthyroidism

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 66 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Central sensitization | 7 days
  The patients will be evaluated for central sensitization with Central Sensitization Inventory. The Central Sensitization Inventory assesses 25 health-related symptoms. Responses are recorded about the frequency of each symptom, with a Likert scale from 0 (never) to 4 (always), resulting in a total possible score of 100. Higher scores are associated with a higher degree of self-reported symptomology.
Headache-related disability | 3 months
  The patients will be evaluated for headache-related disability with The Migraine Disability Assessment Test. Migraine Disability Assessment scores (numerical scores represent number of days patients missed or lost productivity at work or school, as well as missed days from family/social/leisure activities, and range from little or no disability (0-5) to severe disability (>20).
The impact of headache on quality of life | 3 months
  The patients will be evaluated for the impact of headache on quality of life with 6-item short-form Headache Impact Test. This test is a patient-reported outcome measure used to measure the impact and effect of headache on the ability to function normally in daily life. It consists of 6 questions, total scores may range from 36 to 78 and higher scores reflecting greater impact.
Allodynia | 7 days
  The patients will be evaluated for allodynia with the Allodynia Symptom Checklist. The Allodynia Symptom Checklist include 12 questions about the frequency of various allodynia symptoms in association with headache attacks. Instead of using a dichotomous option (yes or no), the response categories are "never," "rarely," "less than half the time," and "half the time or more." In addition, subjects can also indicate that an item "does not apply to me." That option is used by someone who never shaved their face or someone who never wore a ponytail.
Health-Related Quality | 7 days
  The patients will be evaluated for the quality of life with The Short Form-36. This form is composed of 36 items and eight subscales to evaluate quality of life (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health). The scores of the subscales range between 0 and 100, and higher scores indicate higher quality of life.
Sleep quality | 7 days
  The patients will be evaluated for sleep quality with the Pittsburgh Sleep Quality Index. It contains 19 self-reported items and 5 items to be completed by a bed partner or roommate, if possible. Scores range from 0 to 3, and are summed to obtain a global score, which ranges from 0 to 21. Higher scores indicate greater sleep disturbance.
Anxiety and depression | 7 days
  The patients will be evaluated for anxiety and depression with Hospital Anxiety and Depression Scale. The scale is a fourteen-item scale with seven items each for anxiety and depression subscales. Scoring for each item ranges from zero to three. A subscale score >8 denotes anxiety or depression.
The quality of life and functional status of patients with fibromyalgia | 1 month
  The quality of life and functional status of patients with fibromyalgia syndrome will be evaluated with the Fibromyalgia Impact Questionnaire. In this scale, 10 different characteristics are measured, including physical function, well-being, inability to work, difficulty at work, pain, fatigue, morning tiredness, stiffness, anxiety, and depression. The maximum score is 100, and increased score represents decreased functionality.

SECONDARY OUTCOMES:
Descriptive information | 3 months
  Date of birth, education level, body mass index, occupation, marital status, socioeconomic status, age of onset of migraine complaints, descriptive information about migraine attacks (type (with or without aura), duration of attacks, average number of days with pain, pain severity, accompaniments) will be questioned. In addition, if the patient meets the diagnostic criteria of fibromyalgia syndrome, symptom duration and average body pain severity in the last 3 months will be questioned.

CONTACTS AND LOCATIONS:
Overall Officials: Uğur Uygunoğlu, MD, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University- Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No